CLINICAL TRIAL: NCT03720418
Title: A Phase I/II Safety and Dose Evaluation Study of OXB-102 (AXO-Lenti-PD) in Patients With Bilateral Idiopathic Parkinson's Disease (SUNRISE-PD)
Brief Title: Study of OXB-102 (AXO-Lenti-PD) in Patients With Bilateral, Idiopathic Parkinson's Disease
Acronym: SUNRISE-PD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: As a result of termination of development of OXB-102-01, it is no longer possible for Sio to either commence or to continue any related clinical trials.
Sponsor: Sio Gene Therapies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXB-102-01
Record Dates: First submitted 2018-10-16; First posted 2018-10-25 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Gene therapy; OXB-102; AXO-Lenti-PD
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study Part A open-label and Study Part B randomized, double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- OXB-102 Dose Level 1 (Experimental): OXB-102 Dose Level 1 Single Administration (Part A: open-label)
  Interventions: Drug: OXB-102
- OXB-102 Dose Level 2 (Experimental): OXB-102 Dose Level 2 Single Administration (Part A: open-label)
  Interventions: Drug: OXB-102
- OXB-102 Dose Level 3 (Experimental): OXB-102 Dose Level 3 Single Administration (Part A: open-label)
  Interventions: Drug: OXB-102
- OXB-102 Selected Dose (Experimental): Selected Dose of OXB-102 Single Administration (Part B: double-blind)
  Interventions: Drug: OXB-102
- Imitation Surgical Procedure (Sham Comparator): General anesthesia with bilateral skin incisions (Part B: double-blind)
  Interventions: Other: Imitation Surgical Procedure (ISP)

INTERVENTIONS:
Drug: OXB-102 — Neurosurgical delivery of OXB-102 (gene therapy) to the putamen
  Other Names: AXO-Lenti-PD
  Arms: OXB-102 Dose Level 1; OXB-102 Dose Level 2; OXB-102 Dose Level 3; OXB-102 Selected Dose
Other: Imitation Surgical Procedure (ISP) — Participants randomized to the control group in Part B will receive an ISP
  Arms: Imitation Surgical Procedure

SUMMARY:
This study consists of two parts. Part A will evaluate the safety and tolerability of multiple doses of OXB-102 (AXO-Lenti-PD) in participants with Parkinson's disease. Part B will assess the safety and efficacy of the selected dose of OXB-102 in participants with Parkinson's disease.

DETAILED DESCRIPTION:
This study consists of two parts. Part A is an open-label dose-escalation phase in which participants are enrolled in cohorts and will receive one of approximately three escalating doses of OXB-102 (AXO-Lenti-PD). Part B is a randomized, double-blind phase in which participants will be randomized to either an active group receiving the selected dose from Part A, or to a control group receiving an imitation surgical procedure (ISP).

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosed with bilateral idiopathic PD
2. Males/females between 30 and 70 years at the time of surgery
3. Unified Parkinson's Disease Rating Scale (UPDRS) (Part III) score of between 30 and 60 in the "OFF" medication state
4. Presence of motor fluctuations and/or dyskinetic movement
5. Candidate for surgical intervention
6. Hoehn and Yahr (H&Y) Stage 3 or 4 in the "OFF" medication state
7. Stable dosing of PD medication, including L-DOPA, for four weeks prior to screening with Levodopa equivalent daily dose (LEDD) of at least 900 mg

Key Exclusion Criteria:

1. History of psychosis or current treatment with dopamine blocking agents and prior regular exposure to antipsychotic agents
2. History of stereotactic or other surgery for the treatment of PD, including Deep Brain Stimulation (DBS)
3. Participation in a prior cell or gene transfer therapy study
4. Contraindications to use of anaesthesia
5. Current or anticipated treatment with anticoagulant therapy or the use of anticoagulation therapy that cannot be temporarily stopped around the time of surgery
6. Diagnosis of multiple system atrophy
7. Abnormal MRI findings such as mega cisterna, septum pellucidum, signs of severe cortical or subcortical atrophy, brain tumours, vascular diseases, trauma or arteriovenous malformations
8. Presence of dementia

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Safety of OXB-102 as measured by incidence of treatment emergent adverse events and serious adverse events | 3 months timepoint
  Treatment emergent adverse events and serious adverse events will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, for severity
Safety of OXB-102 as measured by changes in clinical laboratory analysis | 3 months timepoint
  Number of clinically significant changes in clinical laboratory analysis
Safety of OXB-102 as measured by changes in vital signs | 3 months timepoint
  Number of clinically significant changes in vital signs
Safety of OXB-102 as measured by changes in brain MRI findings | 3 months timepoint
  Number of clinically significant changes in brain MRI findings
Safety of OXB-102 as measured by changes in physical examination | 3 months timepoint
  Number of clinically significant changes in physical examination

SECONDARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) scores defined in "OFF" and "ON" medication states | Baseline to 6 months
Change in "OFF" time during waking day compared to baseline as assessed by participant diaries | Baseline to 6 months
Change in dyskinesia rating scale score | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Erika De Boever, DDS, PhD, Study Director — Sio Gene Therapies
Locations (3):
- Service de Neurochirurgie, Hôpital Henri Mondor, Créteil, France
- United Kingdom (2):
  - University of Cambridge, Centre for Brain Repair, Cambridge, Cambridgeshire
  - The National Hospital for Neurology and Neurosurgery, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS: 1. GENE THERAPY FOR PARKINSON'S, 2. PHASE 3 STUDY IN FOCUS - INTEC PHARMA'S ACCORDION PILL, 3. CLINICAL TRIALS RESOURCES. J Parkinsons Dis. 2019;9(2):251-264. doi: 10.3233/JPD-199001. No abstract available. PMID 31127735